CLINICAL TRIAL: NCT02793427
Title: Evaluation of Advanced Glycation End Products of Proteins as a Long-term Retrospective Markers of Glycemic Control in a Population of Non-complicated Type 1 Diabetic Children.
Brief Title: Patient With Any Pathology (According to the Appreciation of the Investigator) Which Could Disturb the Participation in the Study
Acronym: AGEDIA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: CHU de Reims (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: PA10007
Record Dates: First submitted 2016-05-27; First posted 2016-06-08 (Estimated); Last update posted 2016-06-09 (Estimated); Status verified 2016-06

CONDITIONS: Type 1 Diabetes in Children

ARMS (2):
- Type 1 diabetes (Experimental)
  Interventions: Biological: blood sample collection
- control (Experimental)
  Interventions: Biological: blood sample collection

INTERVENTIONS:
Biological: blood sample collection

SUMMARY:
The objective of the study is to quantify the products of non-enzymatic glycation of proteins (called AGEs for advanced glycation end-products) in serum of type 1 diabetic patients without clinical complications in order to define the contribution of this markers in the long-term monitoring of glycemic control in these patients. The results will define the criteria for using these new markers in daily clinical practice for the monitoring of these patients

DETAILED DESCRIPTION:
Primary objective : Determine whether AGEs could serve as long-term retrospective indicators of glycemic control of type 1 diabetic patients and determine how to use these markers in a clinical practice for therapeutic purpose and patient monitoring.

For this purpose, it is necessary to determine baseline and pathophysiological ranges of concentrations for serum AGEs and to find a link between AGEs and glycemic control Secondary objectives: (1) Evaluation of the early predictive potential of AGEs for the onset of diabetes complications. (2) Measurement of fructosamine-3-kinase erythrocyte activity and evaluation of its effect on glycemic control in diabetic patients and on the accumulation of AGEs. (3) Ancillary study: development of new methods of evaluation of glycation of serum proteins based on the use of innovative technologies such as vibrational spectroscopy (Raman and infrared).

Protocol design: Cross-sectional and single-center study using a cohort of diabetic children who will be followed over a period of 5 years. Population / patients: 118 children with type 1 diabetes children without clinical complications and 33 non-diabetic children. The group of patients will be stratified on the duration of diabetes: enrolled at the time of the discovery of diabetes or during follow-up of a previously known diabetes. Control subjects will be recruited among siblings of diabetic patients followed at the University Hospital of Reims and among non-diabetic patients treated at the Hospital of Reims for a disease that does not interfere with the protocol, with a matching on age ± 2 years.

Plan of investigation: First phase: after collecting information and informed consent of the child and the holders of parental authority, inclusion of patients achieving blood samples for all children (control and diabetic). For diabetic patients, this blood collection is included in their follow-up. Thus, no additional sample is necessary for the protocol. Second phase: monitoring of diabetic children with blood and urine samples and measurement of skin fluorescence at 5 years after inclusion. No follow-up is planned for control subjects.

Conduct of the study: Inclusion of patients and blood collection. Determination of AGEs (pentosidine, carboxymethyllysine and MG-H1) by high performance liquid chromatography coupled with tandem mass spectrometry by the Laboratory of Biology and Pediatric Research.

Statistical Analyses: Find a link between type 1 diabetes and AGE concentrations and a link between diabetes duration and concentrations of AGE by a Student test.ROC Curves to propose reference values for concentrations of AGE. Find a link between AGE concentrations and HbA1c values by Spearman correlation test and a link between AGE concentrations and HbA1c values (HbA1c <7.5% / 7.5% <HbA1c <8.5% / HbA1c> 8.5%) by a simple linear regression or a Kruskal Wallis test. Find a link between AGE concentrations and magnitudes of change in HbA1c by Spearman correlation test or Pearson.

ELIGIBILITY:
IInclusion criteria : Diabetic patients

* Patient aged 1-18 years recruited according to the duration of diabetes
* Patient with type 1 diabetes
* Patient without clinical diabetes complications
* Patient and his parents have agreed and signed the informed consent for participation

Control subjects

* Control subjects recruited among the siblings of all diabetes patients followed at the University Hospital of Reims.
* Non-diabetic patient followed at Reims University Hospital for a disease which, according to the appreciation of the investigator, may not interfere with the current protocol and the expected results.
* Obtaining informed consent from the Patient and from the holder of parental authority.

Exclusion criteria : Diabetic patients

* Patient with a monogenic diabetes or MODY diabetes who does not require permanent insulin therapy.
* Patient with any pathology (according to the appreciation of the investigator) which could disturb the participation in the study

Control subjects

* Control subject requiring long-term or frequently corticosteroid treatment or any treatment that may disturb glucose metabolism
* Control subject with chronic disease or a history of severe disease (malignant disease, kidney or liver disease, ...)
* Control subject with significant ongoing or recovering acute disease
* Control subject with obesity (BMI greater than the 97th percentile compared to the reference curves of the evolution of BMI according to age).

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 160 (Estimated)
Dates: Start 2011-02; Primary Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
Serum AGEs | 5 years after the inclusion

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Reims, Reims, France, France